CLINICAL TRIAL: NCT00770965
Title: Phase II Single Dose, Randomized, Double-blind, Multi-center, Parallel-group, Placebo-controlled Study to Assess the Efficacy of Three Dose Levels of AIN457 in Patients With Chronic Plaque-type Psoriasis
Brief Title: Phase II Efficacy Study Looking at a Single-dose of One of Three Dose Levels of AIN457 in Patients With Chronic Plaque-type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2204
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Plaque psoriasis, skin condition, thickening, flaking, skin disease, autoimmune disease
MeSH Terms: conditions — Skin Diseases; Autoimmune Diseases | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AIN457 0.3 mg/kg (Experimental): Participants received AIN457 0.3 mg/kg IV on Day 1.
  Interventions: Biological: AIN457
- AIN457 1.0 mg/kg (Experimental): Participants received AIN457 1.0 mg/kg IV on Day 1.
  Interventions: Biological: AIN457
- AIN457 3.0 mg/kg (Experimental): Participants received AIN457 3.0 mg/kg IV on Day 1.
  Interventions: Biological: AIN457
- Placebo (Placebo Comparator): Participants received placebo to AIN457A IV on day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AIN457
  Arms: AIN457 0.3 mg/kg; AIN457 1.0 mg/kg; AIN457 3.0 mg/kg
Biological: Placebo
  Arms: Placebo

SUMMARY:
This is an exploratory, 4 arm, parallel group, placebo-controlled study comparing three doses of AIN457 to placebo. Subjects with a diagnosis of moderate to severe chronic plaque psoriasis will be randomized to receive either AIN457 at one of the three doses studied or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis for at least 6 months prior to screening. The patients must meet all of the following criterion:

  1. Coverage of the body surface area (BSA) of 10% or more with plaques
  2. A score of 3 or more on the IGA (Investigator Global Assessment) scale
  3. A PASI score of at least 12 at baseline;

     Exclusion Criteria:
* Have forms of psoriasis other than the required "plaque psoriasis"
* Women of childbearing potential
* Recent use of investigational drugs or treatment with other biological therapies (wash-out periods required)
* Previous treatment with this investigational drug
* Subjects with active or history of clinically significant cardiac, kidney or liver abnormalities

Other protocol-defined inclusion/exclusion criteria may have applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09-10 (Actual); Primary Completion 2009-09-17 (Actual); Study Completion 2009-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 participants were enrolled into the study. However, due to audit findings at one site, all 65 participants enrolled at the site were excluded from the planned efficacy analyses. As a result, efficacy could not be analyzed due to an insufficient number of participants. The safety set included participants from all other sites.
Period: Safety Set
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo
Started | 2 | 4 | 4 | 5
Completed | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Period: Excluded Set
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo
Started | 18 | 16 | 16 | 15
Completed | 3 | 3 | 2 | 2
Not Completed | 15 | 13 | 14 | 13
Not completed — Administrative problems | 14 | 12 | 12 | 10
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 2 | 4 | 4 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (9.19) | 53.3 (11.79) | 51.5 (8.35) | 52.4 (14.05) | 52.5 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 3 | 7
  Male | 1 | 2 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: This study was not powered for efficacy. Due to audit findings at one site, which included 65 participants, all participants enrolled at the site were excluded from the planned efficacy analyses. As a result, efficacy could not be analyzed due to an insufficient number of participants.
Time Frame: baseline, week 4
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in PASI
Description: This study was not powered for efficacy. Due to audit findings at one site, which included 65 participants, all participants enrolled at site were excluded from the planned efficacy analyses. As a result, efficacy could not be analyzed due to an insufficient number of participants.
Time Frame: baseline, weeks 12, 14, 16, 20, 24, 28 and 32
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Investigator Global Assessment (IGA) Scores
Description: as for outcome 1
Time Frame: baseline, day 1, weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24, 28, 32
Arm/Group | AIN457 0.3 mg/kg | AIN457 1.0 mg/kg | AIN457 3.0 mg/kg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- AIN457 0.3 mg/kg: AIN457 0.3 mg/kg
- AIN457 1 mg/kg: AIN457 1 mg/kg
- AIN457 3 mg/kg: AIN457 3 mg/kg
- Placebo: Placebo
Arm/Group | AIN457 0.3 mg/kg | AIN457 1 mg/kg | AIN457 3 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 4/20 | 5/20 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 0.3 mg/kg (N=20) | AIN457 1 mg/kg (N=20) | AIN457 3 mg/kg (N=20) | Placebo (N=20)
FEMORAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 0.3 mg/kg (N=20) | AIN457 1 mg/kg (N=20) | AIN457 3 mg/kg (N=20) | Placebo (N=20)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
NECROTISING COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CYST (General disorders) | 0 | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0 | 0 | 0
GENITAL HERPES (Infections and infestations) | 0 | 0 | 0 | 1
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 2 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 1
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 2 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.